CLINICAL TRIAL: NCT05558943
Title: Study of Management and Prognosis of Patients With Acute Myeloblastic Leukemia in Saint-Antoine Hospital
Acronym: LAMSA
Status: Not yet recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP211337
Record Dates: First submitted 2022-06-10; First posted 2022-09-28 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-04

CONDITIONS: Acute Myeloid Leukemia
Keywords: Prognosis of Acute myeloblastic leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
AML in adults represents a group of heterogeneous diseases; the prognosis remains poor despite significant therapeutic advances in recent years. In order to optimize patient care, it is necessary to have "real life" data that exhaustively reports on the patients treated in our department. The objective of this study is:

* To describe the AML treated within the hematology department
* To optimize the management of patients with AML.

DETAILED DESCRIPTION:
Current state of knowledge:

Acute myeloblastic leukemia are the most common leukemias in adults. This pathology is very heterogeneous. It has a poor prognosis despite numerous therapeutic advances. The lack of randomized clinical trials can make certain treatment decisions difficult. In addition, patients with comorbidities or the elderly are most often excluded from these trials even though they represent a significant proportion of new diagnoses.

Objectives:

Primary objective Evaluate the overall survival of adult patients treated for AML in our hematology department at Saint-Antoine Hospital.

Secondary objectives

* Evaluate early mortality at 30 days and 60 days post-induction
* Evaluate the CR/CRi rate after induction
* Evaluate the toxicity of the treatments
* Evaluate the relapse-free survival time
* Assess the prognostic value of JC-1 at diagnosis
* Evaluate the proportion of patients eligible for intensive treatment and/or allograft
* Evaluate the side effects of the treatments undertaken
* Describe the molecular and cytogenetic characteristics of hemopathies at diagnosis and at relapse

Duration of study:

Retrospective cohort (cohort A): patients diagnosed between junuary1,2010 and May 30,2022 Prospective cohort (cohort B): patients diagnosed between June 1, 2022 and December 31, 2023. A follow-up of 2 years will be necessary after the end of treatment.

The end of follow-up is estimated at December 2025 for the entire cohort.

Data collection:

Collection of clinical and biological data in the patient's medical file via the Orbis software

Population:

Adult patients treated for AML at Saint-Antoine hospital

ELIGIBILITY:
Inclusion Criteria:

* Age :18 years and older
* Patients with AML
* Non objection to research

Exclusion Criteria:

* Minor patients
* Acute promyelocytic leukemia (AML3)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients treated for AML at Saint-Antoine hospital
Sampling Method: Non-Probability Sample
Enrollment: 750 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2030-06 (Estimated); Study Completion 2030-06 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 2 years after diagnosis

SECONDARY OUTCOMES:
Overall survival | 6 months after diagnosis
Overall survival | 1 year after diagnosis
Cytological remission rate | after the phase of induction up to 24 months
Incomplete cytological remission rate | after the phase of induction up to 24 months
Leukemia free survival rate | 24 months
Side effects | 24 months
  according to the CTCAE v5.0 classification
the rate of patients receiving intensive treatment | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Alexis GENTHON, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Department of Hematology, Hospital Saint Antoine, Paris, France

IPD SHARING:
Plan to Share IPD: No